CLINICAL TRIAL: NCT03276221
Title: Cognitive Recovery With Cannabis Abstinence Among High School-Aged Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Randi Melissa Schuster, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1K23DA042946 (NIH)
Record Dates: First submitted 2017-09-06; First posted 2017-09-08 (Actual); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Cannabis Use; Cognitive Change; Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior | interventions — Natural Family Planning Methods

STUDY DESIGN:
Intervention Model Description: Cannabis users are randomized either to 30 days of cannabis abstinence or 30 days of monitoring with no abstinence requirement. Non-users are not randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Abstinent (Active Comparator): This group of cannabis users are agree to remain abstinent from cannabis use for 30 days.
  Interventions: Behavioral: Abstinence
- Monitoring (No Intervention): This group of cannabis users are not asked to change their cannabis use behavior.
- Non-Users (No Intervention): This is a group of adolescents with little to no cannabis use history and is non-randomized.

INTERVENTIONS:
Behavioral: Abstinence — Cannabis users randomized to this condition will be enrolled in a contingency management intervention for 30 days of cannabis abstinence.
  Other Names: Contingency Management
  Arms: Abstinent

SUMMARY:
This study will use a randomized controlled design to test whether 30 days of cannabis abstinence, compared to 30 days of monitoring, is associated with improvements in cognitive functioning. Non-using controls will also be enrolled to determine the clinical significance of any cognitive improvements with abstinence.

DETAILED DESCRIPTION:
This is a 5-year randomized, longitudinal trial of cannabis abstinence designed to determine (1) if performance improves with abstinence beyond that observed with continued cannabis use, and if so, (2) when during abstinence cognitive improvement occurs, and (3) whether performance in abstinent individuals "returns" to performance levels observed in non-using peers. We hypothesized that abstinent adolescent cannabis users would have more neurocognitive improvement over four weeks compared to non-abstinent cannabis users, and performance would continuously improve throughout four weeks of abstinence. We will recruit 210 adolescents with and without regular cannabis use. Eligible cannabis users will be randomized to either a contingency management intervention which will incentivize 4 weeks of cannabis abstinence (n = 70), or non-contingent monitoring with no abstinence requirement (n = 70). All participants (including non-users; n = 70) will complete cognitive assessments, toxicology testing, self-report questionnaires and semi-structured mood and substance use interviews during the 4-week study as well as one 30-day follow-up visit. Abstinence will be indexed by decreasing levels of cannabis metabolites in urine.

ELIGIBILITY:
General Inclusion Criteria for School-Aged Study Component:

* Male and female adolescents from the Boston area who are between the ages of 10 and 19 (inclusive);
* Have a parent or legal guardian who is able and willing to provide written informed consent for the active study phase (if under the age of 18);
* Competent and willing to provide written informed assent for the active study phase (if under the age of 18);
* Competent and able to provide written informed consent (if age 18 or older)
* Able to communicate in English language
* Able to commit to 9 study visits in approximately 60 days
* No severe developmental delays (including, but not limited to, Autism Spectrum Disorder, Intellectual Disability, and Down Syndrome)
* Able to safely participate in the protocol and appropriate for outpatient level of care

Cannabis-Using Group Inclusion Criteria:

* Use of cannabis at least once per week on most weeks
* Cannabis use reported within 7 days of both baseline visits
* No immediate plan to discontinue cannabis use

Non-Using Group Inclusion Criteria:

* Use of cannabis less than 5 times in lifetime
* No cannabis use in the past year
* No cannabis use before age 16

Exclusion Criteria for School-Aged Study Component

- Passive consent for initial school-wide assessment withdrawn by parent or legal guardian or written parental consent not provided prior to screening

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 201 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2022-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randi M Schuster, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Cooke ME, Gilman JM, Lamberth E, Rychik N, Tervo-Clemmens B, Evins AE, Schuster RM. Assessing Changes in Symptoms of Depression and Anxiety During Four Weeks of Cannabis Abstinence Among Adolescents. Front Psychiatry. 2021 Jul 1;12:689957. doi: 10.3389/fpsyt.2021.689957. eCollection 2021. PMID 34276449
- [Result] Savulich G, Rychik N, Lamberth E, Hareli M, Evins AE, Sahakian BJ, Schuster RM. Sex Differences in Neuropsychological Functioning are Domain-Specific in Adolescent and Young Adult Regular Cannabis Users. J Int Neuropsychol Soc. 2021 Jul;27(6):592-606. doi: 10.1017/S1355617720001435. PMID 34261559
- [Result] Schuster RM, Gilman J, Schoenfeld D, Evenden J, Hareli M, Ulysse C, Nip E, Hanly A, Zhang H, Evins AE. One Month of Cannabis Abstinence in Adolescents and Young Adults Is Associated With Improved Memory. J Clin Psychiatry. 2018 Oct 30;79(6):17m11977. doi: 10.4088/JCP.17m11977. PMID 30408351
- [Result] Schuster RM, Potter K, Lamberth E, Rychik N, Hareli M, Allen S, Broos HC, Mustoe A, Gilman JM, Pachas G, Evins AE. Alcohol substitution during one month of cannabis abstinence among non-treatment seeking youth. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Apr 20;107:110205. doi: 10.1016/j.pnpbp.2020.110205. Epub 2020 Dec 9. PMID 33309538
- [Result] Schuster RM, Potter K, Vandrey R, Hareli M, Gilman J, Schoenfeld D, Evins AE. Urinary 11-nor-9-carboxy-tetrahydrocannabinol elimination in adolescent and young adult cannabis users during one month of sustained and biochemically-verified abstinence. J Psychopharmacol. 2020 Feb;34(2):197-210. doi: 10.1177/0269881119872206. Epub 2019 Sep 19. PMID 31535597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted from 2017 to 2022.
Groups:
- Abstinent: This group of cannabis users agreed to remain abstinent from cannabis use for 30 days.
  Abstinence: Cannabis users randomized to this condition will be enrolled in a contingency management intervention for 30 days of cannabis abstinence.
- Monitoring: This group of cannabis users were not asked to change their cannabis use behavior.
- Non-Users: This is a group of adolescents with little to no cannabis use history and were non-randomized.
Period: Overall Study
Arm/Group | Abstinent | Monitoring | Non-Users
Started | 64 | 68 | 69
Completed | 54 | 66 | 69
Not Completed | 10 | 2 | 0
Not completed — Lost to Follow-up | 6 | 2 | 0
Not completed — Did not abstain from cannabis as per protocol | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abstinent | Monitoring | Non-Users | Total
Number analyzed (Participants) | 54 | 66 | 69 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.3 (1.4) | 18.1 (1.5) | 17.0 (1.8) | 17.8 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 31 | 40 | 97
  Male | 28 | 35 | 29 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 16 | 9 | 30
  Not Hispanic or Latino | 49 | 50 | 60 | 159
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 4 | 7 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 10 | 14 | 34
  White | 31 | 34 | 39 | 104
  More than one race | 6 | 11 | 4 | 21
  Unknown or Not Reported | 2 | 3 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 54 | 66 | 69 | 189
APSS [Mean (Standard Deviation); unit: Score on a scale] — Adolescent Psychotic Symptom Screener (APSS). Summed score over 7 items ranging from 0 to 7, where higher scores indicate more psychotic symptoms.
  Score on a scale | 0.1 (0.6) | 0.3 (0.8) | 0.1 (0.5) | 0.2 (0.7)
PQB [Mean (Standard Deviation); unit: Score on a scale] — Prodromal Questionnaire- Brief (PQB). Summed score of 21 items ranging from 0 to 21, where higher scores indicate more prodromal symptoms.
  Score on a scale | 2.9 (3.7) | 3.8 (3.8) | 1.8 (2.3) | 2.8 (3.4)
Years Spent Using Cannabis [Mean (Standard Deviation); unit: years] | 3.3 (1.3) | 3.4 (1.5) | 0 (0) | 3.4 (1.4)
Days Per Month Spent Using Cannabis [Mean (Standard Deviation); unit: days] | 3.6 (2.8) | 3.3 (2.6) | 0 (0) | 3.5 (2.7)
THC-COOH [Mean (Standard Deviation); unit: ng/mL] | 211.8 (338) | 389.6 (745) | 0 (0) | 306.3 (594.6)
CUDIT-R [Mean (Standard Deviation); unit: Score on a scale] — Cannabis Use Disorder Identification Test - Revised (CUDIT-R). Summed score over 8 items ranging from 0 to 32, where higher scores indicate more problematic cannabis usage.
  Score on a scale | 13.7 (5.4) | 14.1 (5.5) | 0 (0) | 13.9 (5.4)
Days Per Month Spent Drinking Alcohol [Mean (Standard Deviation); unit: days] | 0.7 (0.8) | 0.4 (0.8) | 0.1 (0.2) | 0.4 (0.7)
AUDIT [Mean (Standard Deviation); unit: Score on a scale] — Alcohol Use Disorder Identification Test (AUDIT). Summed score over 10 items ranging from 0 to 40, where higher scores indicate more problematic alcohol usage.
  Score on a scale | 5.4 (4.8) | 5.9 (5.0) | 1.9 (2.5) | 4.3 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in the Total Number of Errors From Paired Associates Learning (PAL) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The number of times the subject chose the incorrect box for a stimulus on assessment problems plus an adjustment for the estimated number of errors they would have made on any problems/attempts/recalls they did not reach. This is a specific measure from the Paired Associates Learning (PAL) module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The PAL module assesses visual memory and new learning. Count variable, ranging from 0 to 70, where higher scores indicate more errors and worse performance.
Time Frame: 1, 2, 3, and 4 Weeks
Population: Pre-specified confirmatory analyses assessed differences between the abstinent and monitoring arms only (see attached Statistical Plan).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 5.6 (6.4) | 6.2 (7.7) | 5.9 (8.1)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; The mean difference in scale scores between the abstinence and monitoring groups was estimated via a binomial model with a dummy-coded contrast (0 for monitoring, 1 for abstinence). The model adjusted for change at weeks 2, 3, and 4 of the study, and for a subject's scale scores at baseline; Test type: Superiority; p = 0.215, Mixed Models Analysis — The p-value was adjusted for multiple comparisons by the Bonferroni correction across outcomes for the paired associates learning module. The a priori threshold for statistical significance was 0.025; Estimates were obtained using generalized estimating equations (GEE) with robust standard errors obtained by the sandwich estimator; Slope = -0.19, Standard Error of Mean 0.15 — The estimate is the mean difference in the log probability of making an error for the abstinence group above and beyond the monitoring group (positive values indicate higher error commission for the abstinence group)

2. Primary Outcome: Mean Difference in First Attempt Memory Score From Paired Associates Learning (PAL) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The number of times a subject chose the correct box on their first attempt when recalling pattern locations, which was calculated across all trials. This is a specific measure from the Paired Associates Learning (PAL) module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The PAL module assesses visual memory and new learning. Count variable, ranging from 0 to 20, where higher scores indicate better memory performance.
Time Frame: 1, 2, 3, and 4 Weeks
Population: Pre-specified confirmatory analyses assessed differences between the abstinent and monitoring arms only (see attached Statistical Analysis Plan).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 16.2 (3.2) | 15.8 (3.4) | 16.1 (3.6)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.495, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = 0.10, Standard Error of Mean 0.14 — The estimate is the mean difference in the log probability of picking the correct box for the abstinence group above and beyond the monitoring group (positive values indicate better memory performance for the abstinence group)

3. Primary Outcome: Mean Difference in Forward Span Length From Spatial Span (SSP) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The longest length of sequences (spans) a subject successfully remembered in the original order. This is a specific measure from the Spatial Span (SSP) Module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The SSP assesses visuospatial working memory capacity. Count variable, ranging from 2 to 9, with higher scores indicating better memory performance.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 7.6 (1.3) | 7.4 (1.3) | 7.6 (1.4)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.050, Mixed Models Analysis — The p-value was adjusted for multiple comparisons by the Bonferroni correction across outcomes for the spatial span module. The a priori threshold for statistical significance was 0.025; [statistical method as in outcome 1, analysis 1]; Slope = 0.28, Standard Error of Mean 0.14 — The estimate is the mean difference in the log probability of reaching a longer span for the abstinence group above and beyond the monitoring group (positive values indicate higher span lengths for the abstinence group)

4. Primary Outcome: Mean Difference in Reverse Span Length From Spatial Span (SSP) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The longest length of sequences (spans) a subject successfully remembered in the reverse order. This is a specific measure from the Spatial Span (SSP) Module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The SSP assesses visuospatial working memory capacity. Count variable, ranging from 2 to 9, with higher scores indicating better memory performance.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 6.9 (1.4) | 7 (1.5) | 6.9 (1.6)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.532, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = -0.07, Standard Error of Mean 0.12 — [estimate comment as in outcome 3, analysis 1]

5. Primary Outcome: Mean Difference in the Total Number Correct in the Immediate Recall Measure From the Verbal Recognition Memory (VRM) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The total number of distinct words a subject correctly recalled from the studied list of 18 words during the immediate free recall phase. This is a specific measure from the Verbal Recognition Memory (VRM) Module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The VRM module assesses verbal memory and new learning. Count variable, ranging from 0 to 18, with higher scores indicating better immediate recall performance.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 7.3 (2.3) | 7.3 (2.5) | 7.7 (2.7)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.226, Mixed Models Analysis — The p-value was adjusted for multiple comparisons by the Bonferroni correction across outcomes for the verbal recognition memory module. The a priori threshold for statistical significance was 0.0125; [statistical method as in outcome 1, analysis 1]; Slope = 0.09, Standard Error of Mean 0.07 — The estimate is the mean difference in the log probability of making a correct choice for the abstinence group above and beyond the monitoring group (positive values indicate higher memory performance for the abstinence group)

6. Primary Outcome: Mean Difference in the Total Number Correct in the Delayed Recall Measure From the Verbal Recognition Memory (VRM) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The total number of distinct words a subject correctly recalled from the studied list of 18 words during the delayed free recall phase. This is a specific measure from the Verbal Recognition Memory (VRM) Module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The VRM module assesses verbal memory and new learning. Count variable, ranging from 0 to 18, with higher scores indicating better immediate recall performance.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 6.5 (2.8) | 6.5 (3) | 7.2 (3.1)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.369, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = 0.08, Standard Error of Mean 0.09 — [estimate comment as in outcome 5, analysis 1]

7. Primary Outcome: Mean Difference in the Total Number Correct in the Immediate Recognition Condition From the Verbal Recognition Memory (VRM) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The total number of words a subject correctly identified as either previously studied or novel during the immediate recognition phase. This is a specific measure from the Verbal Recognition Memory (VRM) Module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The VRM module assesses verbal memory and new learning. Count variable, ranging from 0 to 36, with higher scores indicating better recognition memory performance.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 32.3 (2.1) | 32.4 (2.9) | 31.9 (3.1)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.647, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = 0.05, Standard Error of Mean 0.11 — [estimate comment as in outcome 5, analysis 1]

8. Primary Outcome: Mean Difference in the Total Number Correct in the Delayed Recognition Condition From the Verbal Recognition Memory (VRM) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The total number of words a subject correctly identified as either previously studied or novel during the delayed recognition phase. This is a specific measure from the Verbal Recognition Memory (VRM) Module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The VRM module assesses verbal memory and new learning. Count variable, ranging from 0 to 36, with higher scores indicating better recognition memory performance.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 30.5 (3) | 30.9 (3.6) | 30.3 (4)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.511, Mixed Models Analysis — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = -0.06, Standard Error of Mean 0.09 — [estimate comment as in outcome 5, analysis 1]

9. Primary Outcome: Mean Difference in the Total Number Incorrect From the Multitasking Test (MTT) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The total number of words a subject correctly identified as either previously studied or novel during the delayed recognition phase. This is a specific measure from the Multitasking Test (MTT) module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The MTT assesses the participant's ability to manage conflicting information provided by the direction of an arrow and its location on the screen and to ignore task-irrelevant information. Count variable, ranging from 0 to 160, with higher scores indicating more errors and worse performance.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 7.1 (5.6) | 8.5 (7.7) | 9.1 (8.1)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.312, Mixed Models Analysis — The p-value was adjusted for multiple comparisons by the Bonferroni correction across outcomes for the multitasking test module. The a priori threshold for statistical significance was 0.0125; [statistical method as in outcome 1, analysis 1]; Slope = -0.12, Standard Error of Mean 0.12 — [estimate comment as in outcome 1, analysis 1]

10. Primary Outcome: Mean Difference in the Response Latency From the Multitasking Test (MTT) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The response latency for each participant was defined as a summary (median) computed over their response times for all correct responses irrespective of condition. This is a specific measure from the Multitasking Test (MTT) module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The MTT assesses the participant's ability to manage conflicting information provided by the direction of an arrow and its location on the screen and to ignore task-irrelevant information. Response time variable in milliseconds (ms), ranging from 100 to 2000 ms, with higher values indicating slower performance across all trials.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 474 (72) | 468 (78) | 482 (86)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.836, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = 1.92, Standard Error of Mean 9.27 — The estimate is the mean difference in the median response latency for the abstinence group above and beyond the monitoring group (positive values indicate higher slower responses for the abstinence group)

11. Primary Outcome: Mean Difference in the Incongruency Cost From the Multitasking Test (MTT) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The incongruency cost for each participant was defined as a summary (median) of response times for incongruent trials minus a summary (median) of response times for congruent trials. This is a specific measure from the Multitasking Test (MTT) module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The MTT assesses the participant's ability to manage conflicting information provided by the direction of an arrow and its location on the screen and to ignore task-irrelevant information. Difference score in milliseconds (ms), ranging from -1900 to 1900 ms, with higher values indicating slower responses on incongruent trials, suggesting that it takes longer to process conflicting information.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 37 (33) | 40 (32) | 43 (37)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.898, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = -0.50, Standard Error of Mean 3.93 — The estimate is the mean difference in the median incongruency cost for the abstinence group above and beyond the monitoring group (positive values indicate higher costs for incongruent trials for the abstinence group)

12. Primary Outcome: Mean Difference in the Multitasking Cost From the Multitasking Test (MTT) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The multitasking cost for each participant was defined as a summary (median) of response times for the multi-task blocks (trials alternated between having to respond to the direction or position of the arrow) minus a summary (median) of response times for the single-task blocks (all trials consisted of either responding to the direction or position of the arrow). This is a specific measure from the Multitasking Test (MTT) module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The MTT assesses the participant's ability to manage conflicting information provided by the direction of an arrow and its location on the screen and to ignore task-irrelevant information. Difference score in milliseconds (ms), ranging from -1900 to 1900 ms, with higher values indicating slower responses on multi-task blocks, suggesting that it takes longer to process multiple sources of information.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 96 (71) | 71 (68) | 81 (81)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.068, Mixed Models Analysis — [p-value comment as in outcome 9, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = 16.54, Standard Error of Mean 9.05 — The estimate is the mean difference in the multitasking cost for the abstinence group above and beyond the monitoring group (positive values indicate higher costs for multitasking trials for the abstinence group)

13. Primary Outcome: Mean Difference in Number of Problems Correctly Solved on the First Choice From the One Touch Stockings of Cambridge (OTS) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The total number of trials where the subject chose the correct answer on the first attempt. This is a specific measure from the One Touch Stockings of Cambridge (OTS) Module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The OTS module assesses executive function based upon the Tower of Hanoi test. Count variable, ranging from 0 to 15, with higher scores indicating better performance.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 12.2 (1.8) | 11.5 (2.3) | 11.5 (2.7)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.150, Mixed Models Analysis — The p-value was adjusted for multiple comparisons by the Bonferroni correction across outcomes for the one touch stockings of Cambridge module. The a priori threshold for statistical significance was 0.025; [statistical method as in outcome 1, analysis 1]; Slope = 0.15, Standard Error of Mean 0.10 — The estimate is the mean difference in the log probability of making a correct response for the abstinence group above and beyond the monitoring group (positive values indicate higher accuracy for the abstinence group)

14. Primary Outcome: Mean Difference in the Latency to First Correct Choice From the One Touch Stockings of Cambridge (OTS) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The latency to first correct choice for each participant was defined as a summary (median) of the response times for all trials in which the subject picked the correct choice on the first attempt. This is a specific measure from the One Touch Stockings of Cambridge (OTS) Module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The OTS module assesses executive function based upon the Tower of Hanoi test. Response time variable in milliseconds (ms), a positive unbounded variable, with higher values indicating slower performance across correct trials.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 7036 (2794) | 6690 (2283) | 6851 (3183)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.525, Mixed Models Analysis — [p-value comment as in outcome 13, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = 179.11, Standard Error of Mean 281.76 — [estimate comment as in outcome 1, analysis 1]

15. Primary Outcome: Mean Difference in Stop Signal Reaction Time From Stop Signal Task (SST) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The estimate of the duration at which a person can successfully inhibit a response 50% of the time, represents the time before which all actions become ballistic and a subject is unable to cancel a response selection. This is a specific measure from the Stop Signal Task (SST) Module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The SST module assesses response inhibition (impulse control). Response time variable in milliseconds (ms), ranging from 0 to 500 ms, with higher values indicating that it takes longer for a person to inhibit a response.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 210 (35) | 219 (49) | 222 (56)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.038, Mixed Models Analysis — The p-value was adjusted for multiple comparisons by the Bonferroni correction across outcomes for the stop signal task module. The a priori threshold for statistical significance was 0.05; [statistical method as in outcome 1, analysis 1]; Slope = -10.86, Standard Error of Mean 5.24 — The estimate is the mean difference in the inhibition latency for the abstinence group above and beyond the monitoring group (positive values indicate slower inhibition for the abstinence group)

16. Primary Outcome: Mean Difference in the Total Number of Between Errors From the Spatial Working Memory (SWM) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The number of times a subject incorrectly revisited a box that had contained a token in a previous trial across the 4, 6, and 8 box conditions. This is a specific measure from the Spatial Working Memory (SWM) module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The SWM module provides a measure of strategy as well as working memory errors. Count variable, ranging from 0 to 63, with higher scores indicating worse performance.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 3.6 (5.4) | 4.6 (6.3) | 5.5 (7.7)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.576, Mixed Models Analysis — The p-value was adjusted for multiple comparisons by the Bonferroni correction across outcomes for the spatial working memory module. The a priori threshold for statistical significance was 0.025; [statistical method as in outcome 1, analysis 1]; Slope = -0.10, Standard Error of Mean 0.17 — [estimate comment as in outcome 1, analysis 1]

17. Primary Outcome: Mean Difference in the Participant's Strategy for 6-8 Box Conditions From the Spatial Working Memory (SWM) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The number of times subjects began a new search from the same box they started on in previous trials. It is assumed that a person who begins from the same box each time is using a planned strategy to find the tokens. This is a specific measure from the Spatial Working Memory (SWM) module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The SWM module provides a measure of strategy as well as working memory errors. Count variable, ranging from 2 to 14, with higher scores indicating low strategy, meaning a subject began searches from many different boxes.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 5.4 (2.6) | 5.7 (2.6) | 6.1 (2.7)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.296, Mixed Models Analysis — [p-value comment as in outcome 16, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = -0.15, Standard Error of Mean 0.15 — The estimate is the mean difference in the log probability of trials with strategic responding for the abstinence group above and beyond the monitoring group (positive values indicate higher rates of strategic responding for the abstinence group)

18. Secondary Outcome: Mean Difference in the Measure of Discriminability - A' From the Rapid Visual Information Processing (RVP) Module Averaged Over Weeks 1, 2, 3, and 4
Description: A transformation of the proportion of hits and false alarms, providing an estimate of a subject's ability to detect the target sequences of digits after controlling for response bias (i.e., biases to respond or not respond irrespective of the stimuli on screen). This is a specific measure from the Rapid Visual Information Processing (RVP) module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The RVP module assesses sustained attention. Bounded continuous variable, ranging from 0 to 1, where higher scores indicate a greater ability to discriminate between targets and distractors.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 0.94 (0.05) | 0.93 (0.06) | 0.92 (0.08)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.650, Mixed Models Analysis — The p-value was adjusted for multiple comparisons by the Bonferroni correction across outcomes for the rapid visual information processing module. The a priori threshold for statistical significance was 0.025; [statistical method as in outcome 1, analysis 1]; Slope = 0.00, Standard Error of Mean 0.01 — The estimate is the mean difference in the discriminability measure for the abstinence group above and beyond the monitoring group (positive values indicate higher discriminability rates for the abstinence group)

19. Secondary Outcome: Mean Difference in the Reponse Latency for Hits From the Rapid Visual Information Processing (RVP) Module Averaged Over Weeks 1, 2, 3, and 4
Description: The response latency for hits for each participant was defined as a summary (median) over the set of response times for all correct responses (identification of target 3-digit sequences). This is a specific measure from the Rapid Visual Information Processing (RVP) module, which is part of the Cambridge Neuropsychological Test Automated Battery (CANTAB). The RVP module assesses sustained attention. Response time variable in milliseconds (ms), ranging from 100 to 1900 ms, with higher values indicating slower performance in detecting targets.
Time Frame: 1, 2, 3, and 4 Weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abstinent | Monitoring | Non-Users
Number analyzed (Participants) | 54 | 66 | 69
score on a scale | 422 (51) | 428 (97) | 428 (78)
Statistical Analysis 1: Comparison: Abstinent vs Monitoring; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.223, Mixed Models Analysis — [p-value comment as in outcome 18, analysis 1]; [statistical method as in outcome 1, analysis 1]; Slope = -11.64, Standard Error of Mean 9.55 — The estimate is the mean difference in the median response latency for the abstinence group above and beyond the monitoring group (positive values indicate slower responses for the abstinence group)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 60 days.
Description: Adverse events were collected via systematic assessment. Adverse events were collected at each visit from the time the subject provided informed consent up to and including the last study visit using a standardized questionnaire. All adverse events volunteered, observed, or solicited were recorded in the adverse events CRF. Adverse events were recorded with the date of the event, event description, severity, expectedness, and assessment of relationship to study procedures.
Arm/Group | Abstinent | Monitoring | Non-Users
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/66 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/66 | 0/69
Other Adverse Events (participants affected / at risk) | 49/54 | 46/66 | 31/69
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abstinent (N=54) | Monitoring (N=66) | Non-Users (N=69)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 5 (6) | 1 (1)
General disorders (General disorders) | 45 (92) | 34 (50) | 21 (25)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 1 (1) | 6 (7) | 2 (2)
Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (6) | 1 (1)
Psychiatric Disorders (Psychiatric disorders) | 26 (35) | 11 (11) | 6 (9)
Respiratory, Thoracic and Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7) | 7 (7)

LIMITATIONS AND CAVEATS:
Due to the constraints of the COVID-19 pandemic, approximately 6% of all study visits were conducted virtually. Visits were conducted remotely for one of the following reasons: the study site was closed due to hospital policy, the participant tested positive for COVID-19, or they endorsed a COVID-19-related symptom before the study visit. We believe this is a minor limitation of our study since administering the cognitive assessments virtually could have affected data collection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/21/NCT03276221/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT03276221/SAP_001.pdf
  • Informed Consent Form (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/21/NCT03276221/ICF_002.pdf